CLINICAL TRIAL: NCT05794685
Title: The Analgesic Efficacy of Ultrasound Guided Adductor Canal Block Versus 4 in 1 Block in Patients Undergoing Knee Surgeries: A Comparative Randomized Double Blinded Study .
Acronym: No acronym
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Hussein Bahr (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Hussein Bahr, Associated Professor of Anesthesiology and Surgical Intensive Care and pain medicine, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/12022023/saad
Record Dates: First submitted 2023-03-02; First posted 2023-04-03 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Comparing the Analgesic Outcome by ( 4 in 1 Block ) & ( Adductor Canal Block )
Keywords: ultrasound guided adductor canal block .; 4 in 1 block .; knee surgeries .

STUDY DESIGN:
Intervention Model Description: Comparative Randomized Study between 2 groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adductor canal block (Active Comparator): adductor canal block : patients will receive an injection of 30 ml of .25% of Bupivacaine including 4mg of dexamethasone at a point anterior to the femoral artery, deep to the sartorius muscle
  Interventions: Procedure: adductor canal block; Procedure: 4 in one block
- 4 in one block (Active Comparator): 4 in one block : patients will receive an injection of 30 ml of .25% of Bupivacaine including 4mg dexamethasone at the adductor hiatus where the descending genicular artery branches from superficial femoral artery .
  Interventions: Procedure: adductor canal block; Procedure: 4 in one block

INTERVENTIONS:
Procedure: adductor canal block — patients will receive an injection of 30 ml of .25% of Bupivacaine including 4mg of dexamethasone at a point anterior to the femoral artery, deep to the sartorius muscle (adductor canal block).
Procedure: 4 in one block — patients will receive an injection of 30 ml of .25% of Bupivacaine including 4mg dexamethasone at the adductor hiatus where the descending genicular artery branches from superficial femoral artery (4 in one block).

SUMMARY:
Knee surgeries are associated with severe postoperative pain. Improper pain management affects patients' psychological status with prolongation of hospital stay time and rehabilitation period, with the possibility of progression of the acute pain to chronic pain (McCartney CJ, Nelligan K., 2014). Many Pain management options following these surgeries are available: non-opioid analgesics, opioids and regional anesthesia techniques (epidural and peripheral nerve block). Multi-modal analgesia is considered the best option for pain management in knee surgeries. As non-opioid analgesics alone are not effective enough while opioids alone are associated with many risk factors: nausea, vomiting, decrease intestinal motility and respiratory depression with possibility of addiction (Goode VM, Morgan B, et al, 2019)

DETAILED DESCRIPTION:
Knee surgeries are associated with severe postoperative pain. Improper pain management affects patients' psychological status with prolongation of hospital stay time and rehabilitation period, with the possibility of progression of the acute pain to chronic pain (McCartney CJ, Nelligan K., 2014). Many Pain management options following these surgeries are available: non-opioid analgesics, opioids and regional anesthesia techniques (epidural and peripheral nerve block). Multi-modal analgesia is considered the best option for pain management in knee surgeries. As non-opioid analgesics alone are not effective enough while opioids alone are associated with many risk factors: nausea, vomiting, decrease intestinal motility and respiratory depression with possibility of addiction (Goode VM, Morgan B, et al, 2019). Regarding the functional anatomy of the nerve supply to knee joint: The knee is innervated by genicular branches from the nerve to vastus medialis, saphenous nerve, sciatic nerve and the posterior division of obturator nerve. The skin around the knee is supplied by the cutaneous branches from the femoral nerve and the saphenous nerve (Ritesh Roy, Gaurav Agarwal, et al, 2018). The widespread use of ultrasound to advance peripheral nerve block techniques over the past decade has led to enormous growth in the utilization and efficiency of regional anesthesia (Cozowicz, Crispiana & Poeran, et al, 2015). The adductor canal block (ACB) is an interfascial plane block performed in the middle third of the medial side of the thigh. The adductor canal bounded anteriorly by the sartorius muscle, posteriorly and medially by the adductor longus and magnus muscles, and laterally by the vastus medialis muscle. It contains the femoral vein and artery, the saphenous nerve and the nerve to the vastus medialis, both are sensory branches of the femoral nerve. In some individuals, the obturator sensory branch (also a femoral nerve branch) can be affected by local anesthetic infiltration into this area. It can be noted that this block affect sensory branches and avoid blocking the majority of motor branches. The block is most commonly performed using ultrasound guidance (Thiayagarajan MK, Kumar SV,et al 2019). Ultrasound guided 4-in-1 block technique: a new single injection technique described by Roy R, Agarwal G, et al, 2018 for the combined 4 nerves (saphenous nerve, obturator nerve, nerve to vastus medialis and sciatic nerve) with a single injection point is located at the adductor hiatus where descending genicular artery branches from superficial femoral artery. Bupivacaine is a long-acting amide local anesthetic (max. dose 2.5 mg/kg). Symptoms contributed to local anesthetic toxicity include tinnitus, perioral tingling, visual disturbances and dizziness (Shafiei FT, McAllister RK, Lopez J, 2022)

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* ASA grade 1 and 2.
* Age group between 20-60 years.
* Patients who will undergo knee surgeries under neuroaxial anesthesia.

Exclusion criteria:

* Patient refusal.
* Patients who are allergic to any of study drugs.
* Absolute contraindication causes to spinal anesthesia due to coagulopathy, severe aortic/mitral stenosis, or active infection at site of injection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score: resting and dynamic . | 6 hours Postoperative
  Postoperative pain score: resting and dynamic pain using NRS at postoperative 6 hours.Numerical rating scales (NRSs) are the simplest and most commonly used scales. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable." The patient picks (verbal version) or draws a circle around (written version) the number that best describes the pain dimension, usually intensity.
Postoperative pain score: resting and dynamic | 12 hours post operative
  Postoperative pain score: resting and dynamic pain using NRS at postoperative 12 hours.
Postoperative pain score: resting and dynamic | 18 hours post operative
  Postoperative pain score: resting and dynamic pain using NRS at postoperative 18 hours.
Postoperative pain score: resting and dynamic | 24 hours post operative.
  Postoperative pain score: resting and dynamic pain using NRS at postoperative 24 hours.

SECONDARY OUTCOMES:
Change of blood pressure . | Intraoperative
  Change of blood pressure (systolic, diastolic, mean pressure): Evaluation of the blood pressure before and 30min after applying the assigned block before receiving anesthesia. Then, we will calculate the change of blood pressure at the two time points.
Change of heart rate . | Intraoperative
  Change of heart rate: Evaluation of the heart rate before and 30 min after applying the assigned block before receiving anesthesia. Then, we will calculate the change of heart rate at the two time-points
Postoperative opioid requirements . | 24 hours post operative
  First time for opioid rescue and total dose in the frist 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine.Beni-suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No